CLINICAL TRIAL: NCT03547986
Title: Evaluation of Adjunctive Procedural Assessments to Diagnose Post Drug-coated Balloon Flow-limiting Dissection and Residual Stenosis When Angiography is Inconclusive
Brief Title: BIO REsponse Adapted Combination Therapy Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C1706
Record Dates: First submitted 2018-05-18; First posted 2018-06-06 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Peripheral Arterial Disease
Keywords: flow-limiting dissection; residual stenosis
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Intervention Model Description: The existing and new diagnostic method are performed on the same patients (paired data)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duplex Ultrasound (DUS) (Experimental): Standard angiography and DUS are performed on the same patients (paired data)
  Interventions: Diagnostic Test: Duplex Ultrasound (DUS)
- IVUS with Intraarterial pressure measurement (IAP) (Experimental): Standard angiography and Intra-Vascular Ultrasound (IVUS) with Intraarterial pressure measurement (IAP) are performed on the same patients (paired data)
  Interventions: Diagnostic Test: IVUS with Intraarterial pressure measurement (IAP) if needed

INTERVENTIONS:
Diagnostic Test: Duplex Ultrasound (DUS) — Occurrence of a flow-limiting dissection or residual stenosis will be assessed by standard angiography and Duplex Ultrasound
  Other Names: Procedural diagnostic with Duplex Ultrasound (DUS)
  Arms: Duplex Ultrasound (DUS)
Diagnostic Test: IVUS with Intraarterial pressure measurement (IAP) if needed — Occurrence of a flow-limiting dissection or residual stenosis will be assessed by standard angiography and Intra-vascular ultrasound associated to Intraarterial pressure measurement if needed
  Other Names: Procedural diagnostic with IVUS and Intraarterial pressure measurement (IAP)
  Arms: IVUS with Intraarterial pressure measurement (IAP)

SUMMARY:
Both drug-coated balloon and stents have been used for a number of years to treat subjects with Peripheral Artery Disease (PAD) and are recognized as very good treatment methods. However, due to a higher risk of blood clot formation, requiring a longer anticoagulant treatment, and the challenge of treating re growth of tissue extending through the metal mesh of the stent, the physicians try to reserve stent placement to situation where it's really needed, in case of flow-limiting vessel dissection or acute re-narrowing.

The purpose of this study is to evaluate the utility of several procedural diagnostic techniques in helping the physicians to better decide whether a stent is needed or not.

The study will also estimate the safety and efficacy of Passeo-18 Lux drug-coated balloon associated to Pulsar 18 bare metal stent when and where needed to treat PAD

DETAILED DESCRIPTION:
The REACT treatment concept aims at minimizing the metal burden, combining Passeo-18 Lux Drug-Coated Balloon (DCB) with Pulsar-18 thin struts bare metal stent, as low as reasonably achievable (ALARA), while benefiting from the antirestenotic properties of Paclitaxel. However, in order to optimally apply this selective stenting approach, it is needed to clearly identify when a stent is indicated. Angiographic images, even with additional projections, are sometimes insufficient to clearly determine if a dissection is flow-limiting and the subsequent stent requirement. There is currently no definition nor validated method to define flow-limiting dissection in the peripheral arteries. Even though it has been widely used, the classification developed by the National Heart, Lung, and Blood Institute to grade coronary artery dissection as A to F19, based on angiographic appearance cannot be extrapolated to peripheral arteries.

Therefore, the purpose of the study is to evaluate the incremental value of several adjunctive procedural assessments to standard angiography to identify flow-limiting dissection and residual stenosis, and better inform the operator on the stent requirement. In addition, the study will evaluate the safety and efficacy of the REACT algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent before any study specific test or procedure and is willing and able to comply with the required follow-up visits and procedures
* Subject has a chronic, symptomatic lower limb ischemia defined as Rutherford categories 2 to 4

Angiographic criteria:

* Single lesion or consecutive single lesions with a healthy segment(s) of ≤ 2cm in-between
* De novo, restenotic or (re)occluded lesion(s) post Percutaneous Transluminal Angioplasty in the native superficial femoral artery (SFA) and or the proximal popliteal artery (PPA)
* Lesion(s) must be located at least 1 cm distal to the profunda femoris artery and at least 3 cm above the knee joint (radiographic joint space)
* Degree of stenosis ≥70% by visual angiographic assessment
* Vessel diameter ≥ 4 and ≤ 7 mm
* Patent inflow artery, free from significant lesion (>50%) as confirmed by angiography. Treatment of the target lesion is acceptable after successful treatment of inflow iliac and/or common femoral artery lesion. The inflow lesion cannot be treated with a DCB or a Drug Eluting Stent
* Patent infrapopliteal and popliteal artery, i.e., single vessel runoff or better with at least one of the three vessels patent (<50% stenosis) to the ankle or foot with no planned intervention

Exclusion Criteria:

* Previously stented target lesion
* Target lesion/ previously treated with drug-coated balloon <12 months prior to enrollment.
* Use of atherectomy, laser or other debulking devices in the target SFA/PPA vessel during the index procedure.
* Failure to cross the target lesion with the guide wire
* Presence of a complication following pre-dilation of target lesion, which in the opinion of the investigator would not allow the procedure to be performed in accordance with the REACT approach
* Presence of aneurysm in the target vessel.
* Prior on planned major amputation (above the ankle) in the target limb
* Acute ischemia and/or acute thrombosis of the target SFA/PPA vessel prior to enrollment.
* Perforation of the target vessel as evidenced by extravasation of contrast media prior to enrollment
* Known hypersensitivity or contraindication to contrast media that, in the opinion of the investigator, cannot be adequately pre-medicated
* Known hypersensitivity/allergy to Paclitaxel or other components of the investigational devices and comparator (e.g., nitinol, amorphous silicon carbide, polymer)
* Known hypersensitivity or contraindication to antiplatelet, anticoagulant, thrombolytic medications that would be administered during the study
* Subject with uncorrected bleeding disorders
* Subject with renal failure
* Life expectancy less than 12 months due to other comorbidities, that in the investigators opinion, could limit subject ability to comply with the study required follow-up visits/procedure and threaten the study scientific integrity
* Pregnant, breast feeding, or plan to become pregnant in the next 12 months.
* Current participation in another investigational drug or device clinical study that has not completed the primary endpoint at the time of enrollment or that upon investigator judgment could clinically interferes with the current study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of duplex ultrasound | during index procedure
  specificity and sensitivity of duplex ultrasound combined to angiography vs angiography alone

SECONDARY OUTCOMES:
diagnostic accuracy of intraarterial pressure measurement | during index procedure
  specificity and sensitivity of intraarterial pressure measurement combined to angiography vs angiography alone
diagnostic accuracy of intraarterial pressure measurement with IVUS | during index procedure
  specificity and sensitivity of intraarterial pressure measurement with IVUS combined to angiography vs angiography alone
Target lesion stenting rate | during index procedure
Number of stents used per target lesion | during index procedure
Average stent length per target lesion | during index procedure
Average target lesion length stented (full, spot) | during index procedure
DCB technical success | during index procedure
  Delivery and successful use of Passeo-18 Lux DCB to the target lesion to achieve a residual stenosis no greater than 30% in the absence of flow-limiting dissection
Stent technical success | during index procedure
  delivery and successful use of Pulsar-18 to the target lesion to achieve a residual stenosis no greater than 30%
Procedural success | during index procedure
  technical success and no MAEs before discharge
Primary Patency | 1, 6 and 12 months post index procedure
  Primary patency is defined as DUS peak systolic velocity ratio (PSVR) ≤2.5 at the target lesion, in the absence of clinically driven Target Lesion Revascularization (cd TLR).
Major Adverse Event (MAE) | 1, 6 and 12 months post index procedure
  Major adverse event (MAE) is defined as device or procedure related death within 30 days post index procedure, major target limb amputation or cd TLR post index procedure
Major Adverse Cardiac Event (MACE) | 1, 6 and 12 months post index procedure
  Major adverse Cardiac event (MACE) is defined as death all causes, myocardial infarction, stroke, death or major amputation
Major Adverse Limb Event (MALE) | 1, 6 and 12 months post index procedure
  Major adverse limb event (MALE) is defined as severe limb ischemia leading to an intervention or major vascular amputation
Clinically driven Target Lesion Revascularization | 1, 6, 12, 24 and 36 months post index procedure
  Clinical Event Committee adjudicated TLR =Any post index procedure surgical or percutaneous intervention to the target lesion plus 5 mm proximal and distal to the stented lesion edge when a stent is used
Major target limb amputation rate | 1, 6, 12, 24 and 36 months post index procedure
all cause of death rate | 1, 6, 12, 24 and 36 months post index procedure
Hemodynamic improvement | 1, 6 and 12 months post index procedure
  change in Ankel Brachial Index at 1, 6 and 12 months post index procedure compared to baseline
Rate of primary sustained clinical improvement | 1, 6 and 12 months post index procedure
  Improvement in Rutherford Classification of at least one category for claudicants and by wound-healing and resting pain resolution for critical limb ischemia as compared to pre-procedure without the need for repeat TLR
Rate of secondary sustained clinical improvement | 1, 6 and 12 months post index procedure
  Improvement in Rutherford Classification of at least one category for claudicants and by wound-healing and resting pain resolution for critical limb ischemia as compared to pre-procedure including the need for repeat TLR
Health Related Quality of Life | baseline, 1, 6 and 12 months post index procedure
  The Euroquol Group 5 dimension quality of life questionnaire (EQ-5D) is a descriptive system comprising 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The results in a 1-digit number expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes patient's health state.
  The EQ Visual Analogue Scale records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement
Walk Impairment | baseline, 1, 6 and 12 months post index procedure
  The Walk Impairment Questionnaire (WIQ) measure measures self-reported walking distance, walking speed, and stair-climbing ability
Resource utilisation | during index procedure, 12 month
  Costs will be evaluated using specific information on resource use

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Principal Investigator — Sint Blasius Hospital Dendermonde, Belgium; Patrice Bibombe Mwipatayi, MD, Principal Investigator — Royal Perth Hospital; Michael Lichtenberg, MD, Principal Investigator — Clinic Arnsberg
Locations (15):
- Royal Perth Hospital, Perth, Western Australia, Australia
- Austria (2):
  - Medical University Graz, Graz
  - Medizinische Universität Wien, Vienna
- Belgium (3):
  - OLV Ziekenhuis, Aalst
  - A.Z. Sint-Blasius, Dendermonde
  - AZ Groeninge, Kortrijk
- France (2):
  - CHU de Nantes, Nantes
  - Hopital Paris Saint Joseph, Paris
- Germany (6):
  - Karolinen-Hospital, Klinikum Arnsberg, Arnsberg
  - Universitäts-Herzzentrum Freiburg • Bad Krozingen, Bad Krozingen
  - SRH Klinikum Karlsbad-Langensteinbach, Biederbach Baden-Wurttemberg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum, Tübingen
  - GRN Hospital, Weinheim
- Hospital General de Guadalajara, Guadalajara, Spain

IPD SHARING:
Plan to Share IPD: No